CLINICAL TRIAL: NCT05269732
Title: The Impact of Treating Postpartum Depression on Infant Emotion Regulation
Brief Title: CBT for Postpartum Depression and Infant Emotion Regulation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIER CBT
Record Dates: First submitted 2022-02-15; First posted 2022-03-08 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to the treatment group (delivered group CBT plus TAU) or the control group (treatment as usual).
Who Masked: Investigator
Masking Description: The principal investigator, outcome assessors and data analysts will be blinded to participant allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (9-week online CBT group) (Experimental): Participants assigned to the treatment group will continue to receive any healthcare they might already be receiving (e.g. family doctor, midwife, Obstetrician/Gynecologist, etc.) and participate in a 9-week group Cognitive Behavioral Therapy (CBT) intervention for Postpartum Depression (PPD) delivered via Zoom by two trained psychologists, social workers, nurses, and/or psychiatrists.
  Interventions: Behavioral: Group Cognitive Behavioural Therapy (CBT)
- Control (treatment as usual) (No Intervention): The control group will receive standard postnatal care from their obstetrician, midwife, and/or family physician

INTERVENTIONS:
Behavioral: Group Cognitive Behavioural Therapy (CBT) — The 9-week group Cognitive Behavioural Therapy (CBT) intervention for Postpartum Depression (PPD) delivered via Zoom by two trained psychologists. This intervention was developed by Dr. Van Lieshout (Principal Investigator) at the Women's Health Concerns Clinic (WHCC) at St. Joseph's Healthcare Hamilton. It was designed to be brief, simple, and applicable to women in community settings. It consists of 9 weekly 2-hour sessions where core CBT skills are learned and practiced each week. The first half of each session is devoted to core CBT content, including cognitive restructuring. The second half is devoted to group discussions co-led by participants on topics relevant to mothers with PPD (e.g., sleep, supports, role transitions). Homework is assigned at each session.
  Arms: Treatment (9-week online CBT group)

SUMMARY:
The primary objective of this study is to determine if online group cognitive behavioral therapy (CBT) for maternal postpartum depression (PPD) added to treatment as usual (TAU) leads to greater improvements in infant emotion regulation (ER) than maternal receipt of TAU alone immediately post-treatment and 6 months later. This study will also aim to determine what mechanisms PPD treatment leads to changes in infant ER.

DETAILED DESCRIPTION:
A prospective, single-blind, parallel randomized controlled trial (1:1 ratio) that includes an experimental (receipt of a 9-week group CBT intervention delivered online plus TAU) and control group (TAU alone) to address our objectives. Participants will have an EPDS score of 10 or more and an infant 3-12 months of age and be recruited from the community. The experimental group will receive a validated 9-week online group cognitive behavioral therapy (CBT) intervention on Zoom plus TAU. The control group will receive TAU alone. In both groups, TAU will consist of regular care from their family doctor, midwife, OB/GYN an/or any other types of care they may be accessing. The trial intervention consists of nine, 2-hour sessions occurring once per week. The first half of each session is devoted to core CBT content, including cognitive restructuring. The second half is devoted to group discussions co-led by participants on topics relevant to mothers with PPD (e.g., sleep, supports, role transitions). Groups will be delivered by two trained psychologists, social workers, nurses, and/or psychiatrists. Primary objective: Determine if online group cognitive behavioural therapy (CBT) for maternal PPD added to treatment as usual (TAU) lead to greater improvements in infant ER than maternal receipt of TAU alone immediately post-treatment and 6 months later. Secondary objective: Determine the putative mechanisms through which PPD treatment leads to changes in infant ER.

ELIGIBILITY:
Inclusion Criteria:

* women 18 years of age or older
* understand and speak English (so that they can participate in the CBT group and complete study measures)
* live in Ontario (the primary WHCC catchment area)
* have an EPDS score of 10 or more
* meets diagnostic criteria for comorbid psychiatric conditions.
* Infants must be between 4-12 months old at enrollment.

Exclusion Criteria:

* bipolar disorder
* a current psychotic disorder
* substance or alcohol use disorder
* antisocial or borderline personality disorder.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Infant Temperament | 6 months
  Infant Behavior Questionnaire-Revised (IBQ-R): The IBQ-R is a 91-item scale with 14 subscales that measure infant temperament. Temperament refers to the ways individuals think, behave, and react and is heavily influenced by the degree to which infants and toddlers can regulate their emotions. The items on the IBQ ask parents to rate the frequency of specific temperament-related behaviors observed over the past week. Items are scored on a scale of 0-7. Mothers will complete the IBQ-R on their infants immediately before treatment, right after treatment, and at 6 months afterward.
Infant emotion regulation | 6 months
  Emotional Regulation (ER) is comprised of biological and behavioural domains best measured with validated physiological, observational and informant reports that assess this phenomenon across the full range of infant functioning. Physiological measures: Medial Pre-frontal complex (mPFC) activity using functional near-infrared spectroscopy will be used to observe infant emotion regulatory patterns.
Maternal Depression | 6 months
  Edinburgh Postnatal Depression Scale (EPDS): The EPDS is the 10-item gold standard measure of maternal depressive symptoms. Scores range from 0-30, with higher scores indicating worse depressive symptoms. Mothers will complete the EPDS immediately before treatment, right after treatment, and at 6 months afterward.
Maternal Anxiety | 6 months
  The Generalized Anxiety Disorder 7-Item Scale (GAD-7) is a self-report scale that taps generalized anxiety disorder, the most common comorbidity of Postpartum Depression (PPD). Scores range from 0-21 with higher scores indicating worse anxiety symptoms. Mothers will complete the GAD-7 immediately before treatment, right after treatment, and at 6 months afterward.

SECONDARY OUTCOMES:
Brain-to-brain Synchrony (fNIRS) | 6 months
  Changes in Mother-Infant Synchrony: Physiological and behavioural synchrony patterns are thought to shape infant ER development and explain how treating PPD may exert its effects on infants. Brain-to-brain Synchrony (fNIRS): The fNIRS pre-scanning technique will be used.
The Face-to-Face Stillage Paradigm (FFSP) | 6 months
  The Face-to-Face Stillage Paradigm (FFSP) will be used to observe infant emotion regulatory patterns.
Parent-Child Early Relational Assessment (PCERA) | 6 months
  Parent-Child Early Relational Assessment (PCERA) will be used to observe infant emotion regulatory patterns.
Epigenetic Analyses | 6 months
  One saliva sample will be taken from infants and from mothers at each study visit will be used for epigenetic analyses. Epigenetic modifications will be used to mediate and assess the effect of early life interactions on development.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Van Lieshout, MD, PHD, Principal Investigator — Mcmaster
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No